CLINICAL TRIAL: NCT06980207
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, MAD Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Oral LPM526000133 Fumarate Capsules (LY03017) in Healthy Adult Subjects.
Brief Title: A Phase 1, MAD Study to Evaluate the Safety, Tolerability and Pharmacokinetics of LY03017
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03017/CT-CHN-103
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Hallucinations and Delusions Associated With Alzheimer's Disease Psychosis; Hallucinations and Delusions Associated With Parkinson Disease Psychosis; Negative Symptoms of Schizophrenia
MeSH Terms: conditions — Hallucinations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY03017 (Experimental): LY03017 will be administrated with multiple doses from 10mg to 40mg on day 1~5
  Interventions: Drug: LY03017
- LY03017-Placebo (Placebo Comparator): Placebo will be administrated with multiple doses on day 1~5.
  Interventions: Drug: LY03017-Placebo

INTERVENTIONS:
Drug: LY03017 — administered orally
  Arms: LY03017
Drug: LY03017-Placebo — administered orally
  Arms: LY03017-Placebo

SUMMARY:
This is a phase 1，randomized, double-blind, placebo-controlled, MAD study to evaluate the safety, tolerability and pharmacokinetics of oral LPM526000133 Fumarate Capsules (LY03017) in healthy adult subjects

DETAILED DESCRIPTION:
Primary:

To assess the safety and tolerability of multiple oral doses of LY03017 in healthy adult subjects.

Secondary:

To assess the pharmacokinetics (PK) of LY03017 after multiple oral doses of LY03017 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject who voluntarily participate and sign the informed consent form.
* Healthy male/female volunteers aged ≥18 and ≤ 45 years.
* Body weight ≥ 50.0 kg for men and ≥ 45.0 kg for women, and body mass index (BMI) ≥18.5 and < 28.0 kg/m2.
* Able to comply with the lifestyle restrictions.

Exclusion Criteria:

* Subject has a history of allergy to any component of the investigational drug or similar drugs, or allergic constitution.
* Subject has a history of clinically significant medical conditions that may interfere with the study results, including but not limited to blood system, circulatory system, digestive system, urinary system, respiratory system, nervous system, immune system, endocrine system, malignant tumors, mental disorders and metabolic disorders.
* Any surgical condition or condition may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a hazard to the subjects.
* Subject has clinically significant abnormalities in vital signs, laboratory tests, and ECGs, such as Pulse < 55 beats/min or > 100 beats/min, Systolic blood pressure < 90 mmHg or ≥140 mmHg, Diastolic blood pressure < 60 mmHg or ≥90 mmHg.

QT interval (QTc) ≥450 ms (Male) or 460 ms (Female) .

* Subject has used any of over-the-counter products within 7 days or prescription medications within 28 days prior to dosing.
* Subject has a history of surgery within 3 months prior to administration, or failure to recover from surgery, or having an expected surgical plan during the trial.
* Subject positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), HIV antibody (HIV-Ab), or syphilis seroreactivity (Trust).
* Subject has a history of alcohol abuse within 1 year or positive alcohol breath test results.
* Subject has a history of substance abuse within 1 year or a positive urine drug screen.
* Subject who has daily smoking of ≥ 5 cigarettes within 3 months.
* Subject who has special requirements for food, cannot comply with the unified diet or have dysphagia.
* Subject who has consumption of special diet (such as grapefruit, chocolate, coffee, xanthine-rich foods/drinks) within 48 hours prior to dosing and/or subject who has excessive daily consumption of tea, coffee, grapefruit juice, caffeinated beverages for nearly 3 months.
* Subject who has participated in other clinical trials within 3 months before administration.
* Subject has used blood products or being blood donor or blood loss within 3 months.
* Pregnant, lactating women, or positive pregnancy test.
* Subject who refusal to contraception, or plan to donate sperm or ovums.
* Subject who has a history of needle or blood faintness.
* Subject directly involved in this clinical trial.
* Poor compliance or other conditions which would make participation in the study unsuitable.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | up to day 9

SECONDARY OUTCOMES:
Maximum observed concentration at steady state (Cmax,ss) of LPM526000133 in plasma | up to day 9
Time to maximum observed concentration at steady state (Tmax,ss) of LPM526000133 in plasma | up to day 9
Minimum observed concentration at steady state (Cmin,ss) of LPM526000133 in plasma | up to day 9
Area Under the Concentration-Time Curve from Time Zero to Tau over a Dosing Interval at Steady State(AUC0-τ,ss）of LPM526000133 in plasma | up to day 9
The area under the concentration-time curve from time zero extrapolated to infinity at steady state (AUC0-∞,ss) of LPM526000133 in plasma | up to day 9
Apparent terminal elimination half-life (t1/2) of LPM526000133 in plasma | up to day 9
Accumulation ratio (Ra) of LPM526000133 in plasma | up to day 9

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China